CLINICAL TRIAL: NCT06974461
Title: Effects of Blood Flow Restriction Training on Muscle Strength and Physical Function in Individuals With Stroke-Related Sarcopenia: A Randomized Controlled Trial
Brief Title: Effects of Blood Flow Restriction Training on Muscle Strength and Physical Function for Stroke-Related Sarcopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20250109003
Record Dates: First submitted 2025-04-01; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia; Chronic Stroke Patients
MeSH Terms: conditions — Sarcopenia | interventions — Walking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BFR Walking Group (Experimental): Participants in this group will receive blood flow restriction (BFR) walking training. The pressure cuffs will be applied to the proximal thighs. Walking sessions will be conducted on a treadmill at 60% of the participant's maximum walking speed, 3 times per week for 6 weeks. The cuff pressure will begin at 50% of each participant's arterial occlusion pressure (AOP), determined via Doppler ultrasound, and progressively increased every two weeks to a maximum of 200 mmHg.
  Interventions: Procedure: Blood Flow Restriction (BFR) Walking
- Sham-BFR Walking Group (Sham Comparator): Participants in this group will receive sham blood flow restriction walking training. Pressure cuffs will be applied to the proximal thighs but only inflated to 20 mmHg, which does not restrict blood flow. Walking sessions will be performed under the same treadmill conditions as the BFR group (60% of maximum walking speed, 3 sessions per week for 6 weeks).
  Interventions: Procedure: Sham Blood Flow Restriction (Sham-BFR) Walking

INTERVENTIONS:
Procedure: Blood Flow Restriction (BFR) Walking — Participants in this group will undergo a supervised treadmill walking program with blood flow restriction (BFR) applied using BFR pressure cuffs. The cuffs are applied to the proximal thighs, and the training pressure starts at 50% of the participant's arterial occlusion pressure (AOP), increasing every two weeks up to 200 mmHg. Walking is performed at 60% of the maximum walking speed, 20 minutes per session, 3 sessions per week for 6 weeks.
  Arms: BFR Walking Group
Procedure: Sham Blood Flow Restriction (Sham-BFR) Walking — Participants in this group will follow the same supervised treadmill walking protocol as the BFR group but with minimal cuff pressure (20 mmHg), which does not restrict blood flow. This simulates the sensation of BFR without physiological impact. The purpose is to serve as a placebo comparator. Walking is performed at 60% of maximum walking speed, 20 minutes per session, 3 sessions per week for 6 weeks.
  Arms: Sham-BFR Walking Group

SUMMARY:
Effects of Blood Flow Restriction Walking on Muscle Strength and Physical Function in Chronic Stroke Patients with Sarcopenia: A Randomized, Sham-Controlled Trial Primary Objective: To evaluate the effects of BFR walking on muscle strength and physical function in chronic stroke patients with sarcopenia, compared to sham-BFR walking.

Secondary Objective: (1) To explore the potential impact of BFR walking on muscle mass and vascular function in chronic stroke patients with sarcopenia. (2) To assess the influence of BFR walking on quality of life in chronic stroke patients with sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic stroke (≥6 months post-stroke)
* Diagnosed with sarcopenia, based on AWGS 2019 criteria

Exclusion Criteria:

* Stroke occurred within the past 6 months
* Resting systolic blood pressure > 200 mmHg
* Resting diastolic blood pressure > 100 mmHg
* Presence of implanted electronic or metallic devices that interfere with blood flow restriction cuffs
* Contraindication to bioelectrical impedance analysis (e.g., pacemaker, ICD)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-12-28 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | baseline (prior to intervention), 6 weeks post-intervention (End), and 6 weeks after the end of the intervention (Follow-up)
  Isometric peak torque of the target muscle groups will be measured during both extension and flexion using an isokinetic dynamometer. The unit of measurement is Newton-meters (Nm). Higher values indicate greater muscle strength.
Motor Function - Fugl-Meyer Assessment (FMA) | baseline (prior to intervention), 6 weeks post-intervention (End), and 6 weeks after the end of the intervention (Follow-up)
  Motor function will be assessed using the Fugl-Meyer Assessment, a validated and widely used scale to evaluate motor recovery, particularly in individuals with neurological impairments such as stroke. The total score ranges from 0 to 226, with higher scores indicating better motor function. The assessment includes subscales for upper extremity, lower extremity, coordination, and reflex activity.
Aerobic Capacity and Endurance - Six-Minute Walk Test (6MWT) | baseline (prior to intervention), 6 weeks post-intervention (End), and 6 weeks after the end of the intervention (Follow-up)
  Aerobic capacity and walking endurance will be measured using the Six-Minute Walk Test. Participants will be instructed to walk as far as possible in six minutes on a flat, straight surface. The total distance walked will be recorded in meters. This test reflects submaximal functional capacity relevant to daily physical activity.
Mobility - Timed Up and Go Test (TUG) | baseline (prior to intervention), 6 weeks post-intervention (End), and 6 weeks after the end of the intervention (Follow-up)
  Functional mobility will be assessed using the Timed Up and Go Test. Participants will be asked to stand up from a chair, walk 3 meters, turn around, return to the chair, and sit down. The total time taken to complete the task will be recorded in seconds. Shorter times reflect better mobility.
Gait Speed - 10-Meter Walk Test (10MWT) | baseline (prior to intervention), 6 weeks post-intervention (End), and 6 weeks after the end of the intervention (Follow-up)
  Gait speed will be assessed using the 10-Meter Walk Test at maximum safe walking speed. Participants will be instructed to walk a total of 10 meters as fast as safely possible. The time taken to walk the middle 6 meters (excluding acceleration and deceleration zones) will be recorded, and gait speed will be calculated in meters per second (m/s). Higher values indicate better fast walking ability.
Five Times Sit-to-Stand Test (FTSTS) | Baseline, Week 6, Week 12
  The Five Times Sit-to-Stand Test measures the time in seconds (s) required for a participant to rise from a standard chair to a full standing position and return to sitting five times consecutively as quickly as possible, with arms crossed over the chest. A stopwatch will be used. Lower times indicate better lower limb function and power.
Handgrip Strength | Baseline, Week 6, Week 12
  Handgrip strength will be measured in kilograms (kg) using a digital hand dynamometer.

SECONDARY OUTCOMES:
Nutritional Status - Mini Nutritional Assessment Short Form (MNA-SF) | baseline (prior to intervention), 6 weeks post-intervention (End), and 6 weeks after the end of the intervention (Follow-up)
  Nutritional status will be evaluated using the Mini Nutritional Assessment - Short Form (MNA-SF), a validated screening tool for identifying malnutrition or risk of malnutrition in older adults. The total score ranges from 0 to 14. Scores ≥12 indicate normal nutritional status, 8-11 at risk, and ≤7 malnourished.
Quality of Life - Sarcopenia and Quality of Life Questionnaire (SarQoL) | baseline (prior to intervention), 6 weeks post-intervention (End), and 6 weeks after the end of the intervention (Follow-up)
  Quality of life related to sarcopenia will be assessed using the Sarcopenia and Quality of Life Questionnaire (SarQoL), a disease-specific instrument for older adults with reduced muscle mass or function. It covers domains such as physical health, mental health, locomotion, and daily activities. Higher scores indicate better quality of life.
Appendicular Skeletal Muscle Mass (ASM) | Baseline, Week 6, Week 12
  ASM will be assessed using bioelectrical impedance analysis (BIA) and reported in kilograms per square meter (kg/m²). This value is calculated as total limb lean mass divided by height squared, following the AWGS 2019 criteria.
Muscle Thickness (MT) | Baseline, Week 6, Week 12
  Muscle thickness will be measured using B-mode ultrasonography with a high-frequency linear probe. Values will be reported in millimeters (mm). The average of three measurements will be used for each muscle. Muscle Thickness of Rectus Femoris and Medial Gastrocnemius.
Pennation Angle | Baseline, Week 6, Week 12
  Pennation angle will be obtained from ultrasound images using ImageJ software. The angle between the muscle fascicles and deep aponeurosis will be measured in degrees (°).
Cross-Sectional Area (CSA) | Baseline, Week 6, Week 12
  CSA will be measured from transverse ultrasound images and reported in square centimeters (cm²). Measurements will be taken at standardized anatomical landmarks.
Echo Intensity (EI) | Baseline, Week 6, Week 12
  Echo intensity will be calculated using grayscale analysis from ultrasound images and reported in arbitrary units (a.u.), based on pixel brightness (0 = black, 255 = white).

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided